CLINICAL TRIAL: NCT05805397
Title: Motivation Skills Training to Enhance Functional Outcomes for People With Schizophrenia
Brief Title: Effectiveness of Motivation Skills Training (MST)
Acronym: MST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alice Saperstein, PhD, Assistant Professor of Medical Psychology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAU8435; 1R34MH129552-01A1 (NIH); 8394-2 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2023-03-21; First posted 2023-04-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Mental Illness; Motivation Skills
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Randomized group assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivation Skills Training (MST) (Experimental): MST is a weekly group-based skills training intervention that aims to improve knowledge about one's level and sources of motivation, the ability to monitor and regulate (understand and manage) motivation so that one can better initiate and sustain goal-directed behavior
  Interventions: Behavioral: Motivation Skills Training
- Healthy Behaviors Control Group (Active Comparator): HBC is a weekly group-based intervention that provides psychoeducation and skills training to help individuals improve physical health
  Interventions: Behavioral: Healthy Behaviors Control Group

INTERVENTIONS:
Behavioral: Motivation Skills Training — Participants will complete a baseline assessment, receive weekly MST sessions in a group format for a duration of 12 weeks, and will then repeat the assessment battery from baseline immediately following treatment completion and 2-months after.
  Other Names: MST
  Arms: Motivation Skills Training (MST)
Behavioral: Healthy Behaviors Control Group — Participants will complete a baseline assessment, receive weekly HBC sessions in a group format for a duration of 12 weeks, and will repeat the assessment battery from baseline immediately following treatment completion and 2-months after.
  Other Names: HBC
  Arms: Healthy Behaviors Control Group

SUMMARY:
This study will take place at four outpatient clinics serving adults with serious mental illness. Informed consent will be obtained from N=80 individuals with a Diagnostic and Statistical Manual of Mental Illnesses (DSM)-5 diagnosis of schizophrenia or schizoaffective disorder meeting inclusion/exclusion criteria to participate in a randomized controlled trial comparing Motivation Skills Training (MST) to a Healthy Behaviors Control (HBC) group. Eligible participants will receive a baseline assessment including sociodemographic and psychosocial assessments, measures of motivation, goal attainment, and quality of life, as well as measures of executive skills, community functioning, and psychiatric symptoms severity. Both MST and HBC will be implemented as once weekly group therapies. The treatment phase is approximately 12-14 weeks. MST will focus on motivation knowledge and self-regulation skills while HBC will focus on physical health and health-related skills.

DETAILED DESCRIPTION:
Schizophrenia is a major public health problem associated with core motivational deficits that are amongst the strongest predictors of impaired functional outcomes. Without motivation, people are unable to maintain their pursuit of employment or educational goals, engage in treatment, and regularly participate in healthy life decisions. Current pharmacological and psychosocial treatments for schizophrenia have demonstrated limited effectiveness for improving this core symptom. Motivation Skills Training (MST) is a novel intervention that addresses this clinical need. The premise of MST is that knowledge about one's level and sources of motivation underlies the ability to regulate (i.e., understand and manage) motivation, and that motivation self-regulation can in turn facilitate task initiation and persistence. By facilitating goal-directed behavior, MST aims to enhance daily functioning and goal attainment in people with schizophrenia. MST teaches people about motivation and how to self-regulate motivation, empowering individuals to become active agents in controlling their own motivation and behavior. This study uses a 2-phase model of intervention testing to establish the feasibility, acceptability and pilot effectiveness of MST for adults ages 18-65 with a schizophrenia spectrum diagnosis. An initial open trial of MST in one outpatient clinic will provide stakeholder input on the acceptability and clinical utility of MST content and format, informing refinements to the treatment manual. A subsequent randomized controlled trial will test the effectiveness of MST versus a Healthy Behaviors Control (HBC) group, both conducted in the context of routine recovery-oriented services.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. DSM-5 Diagnosis of Schizophrenia or Schizoaffective Disorder
3. Medically and psychiatrically stable outpatient status
4. English Fluency

Exclusion Criteria:

1. Indications of Intellectual Disability as documented in medical history or measured by < 70 premorbid full scale Intelligence Quotient (IQ) estimate
2. Severe substance use within the past three months determined by DSM-5 criteria
3. Neurologic condition causing brain disease
4. Mild to severe cognitive impairment associated with possible dementia measured by a Mini Mental Status Exam score below 20 in individuals ages 60 and older

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Motivation and Pleasure Scale (MAP) | 5 months
  MAP is a 9-item interviewer rated measure of motivation, pleasure, and engagement in work, school, recreational and social activities. The MAP total score is the sum of all items with a possible range from 0 to 36, with lower scores indicating better outcomes.
Goal Attainment Scaling (GAS) | 5 months
  GAS measures progress towards personal goal attainment, rated along a continuum of predetermined successful outcomes on a scale from 0 to 10. A single rating is used to quantify goal attainment with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Heinrich's Quality of Life Scale (QLS) | 5 months
  QLS is a semi-structured interview which evaluates psychosocial functional outcome. QLS is scored by summing the 7 items reflecting four domains: interpersonal functioning, intrapsychic foundations, instrumental role function, and common objects/activities. Total scores ranges from 0 to 42 where higher scores indicate better functioning.

OTHER OUTCOMES:
Barkley Deficits in Executive Functioning Scale - Short Form (BDEFS-SF) | 5 months
  BDEFS-SF is a self report measure of executive skills relevant to goal-directed behaviors. A summary score is the sum of all 20 items, each rated on a 4-point scale, with a range of 20 to 80 where higher scores indicate greater severity of executive dysfunction.
Specific Levels of Functioning (SLOF) | 5 months
  SLOF rates functioning with each item scored on a 5-point scale measuring physical functioning, personal care skills, interpersonal relationships, social acceptability, activities of community living, and work skills. Scores within each domain are the sum of all domain items with higher scores reflecting better functioning.
Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCI-PANSS) | 5 months
  SCI-PANSS is a semi-structured interview that assesses symptoms of psychotic disorders. Items are each rated from 1 to 7. The total score is the sum of all items, ranging from 30-210, with higher scores indicating greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Saperstein, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - The Bridge, Inc., New York, New York
  - New York State Office of Mental Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
A list of all data expected to be collected in association with this clinical trial will be submitted to the National Institute of Mental Health (NIMH) Data Archive. Descriptive and raw data will be submitted on a semi-annual basis.
Time Frame: Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion, or when the data are published, whichever is earlier
Access Criteria: All data and materials will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with the NIMH Data Archive.